CLINICAL TRIAL: NCT02625779
Title: A Double-Blind, Placebo-Controlled Trial of Combined Cytidine- and Creatine-containing Drug and Dietary Supplement in the Treatment of the Bipolar Depression
Brief Title: Combined Cytidine and Creatine-containing Drug in the Treatment of the Bipolar Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The research project has been cancelled before any participants were enrolled.
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NARSAD_Bipolar
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Depression, Bipolar
Keywords: Bipolar depression; Cytidine; Creatine; Magnetic resonance spectroscopy
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Cytidine; Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Valproate and Placebo (Active Comparator): Valproate: 300mg/day for 8 weeks Placebo: for 8 weeks
  Interventions: Drug: Valproate and Placebo
- Valproate and Cytidine-containing Drug (Experimental): Valproate: 300mg/day for 8 weeks Cytidine-containing Drug: 2g/day for 8 weeks
  Interventions: Drug: Valproate and Cytidine-containing Drug
- Valproate and Creatine-containing Drug (Experimental): Valproate: 300mg/day for 8 weeks Creatine-containing Drug: 3g/day for the first week 5g/day for week 2-8
  Interventions: Drug: Valproate and Creatine-containing Drug

INTERVENTIONS:
Drug: Valproate and Placebo
  Arms: Valproate and Placebo
Drug: Valproate and Cytidine-containing Drug
  Arms: Valproate and Cytidine-containing Drug
Drug: Valproate and Creatine-containing Drug
  Arms: Valproate and Creatine-containing Drug

SUMMARY:
This research is aimed to investigate the efficacy and safety of the creatine and cytidine augmentation in treating bipolar depression and to evaluate changes in relevant brain biochemical metabolism using proton and phosphorous magnetic resonance spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-65 years
* Bipolar disorder I or II (DSM-IV-TR) with current depressive episode
* Informed consent

Exclusion Criteria:

* Use of medication for bipolar depression or other psychotropic drugs
* Current Axis I mental disorders other than bipolar depression based on structured clinical interview
* Current borderline or antisocial personality disorder based on structured clinical interview
* Major medical or neurological illnesses (epilepsy, multiple sclerosis, brain tumor, cerebrovascular disease, etc)
* Hypersensitivity to divalproate or valpromide
* Diagnosis of porphyria
* Current or past liver diseases
* Severe dysfunction in liver or pancreas
* Use of mefloquine
* Alcohol or substance abuse/dependence
* Intelligence quotient of 80 or below
* Contraindications to magnetic resonance imaging
* Pregnancy or breastfeeding
* Allergy or intolerance to the study drugs

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Estimated); Primary Completion 2017-04-30 (Estimated); Study Completion 2017-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of bipolar depression | Baseline and 8 weeks
  assessed with structured clinical interview
Change in depressive symptoms | Baseline and 8 weeks
  assessed with structured clinical interview

SECONDARY OUTCOMES:
Change in brain Glx (glutamate+glutamine) level | Baseline and 8 weeks
  assessed with proton magnetic resonance spectroscopy
Change in brain phosphocreatine level | Baseline and 8 weeks
  assessed with phosphorous magnetic resonance spectroscopy
Number of participants with adverse events | Baseline through 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea